CLINICAL TRIAL: NCT03521869
Title: The Need for Compression Bandage Following Total Knee Arthroplasty A Prospective Randomized Controlled Trial Conducted in Simultaneous Bilateral Total Knee Replacements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14WHoz
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Compression Bandages

STUDY DESIGN:
Intervention Model Description: Only bilateral knee replacements will be utilized so each patient can serve as their internal control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Compression bandage group (Active Comparator)
  Interventions: Device: Compression bandage
- Standard gauze group (Active Comparator)
  Interventions: Device: Gauze dressing

INTERVENTIONS:
Device: Compression bandage — Compression bandage placed after total knee replacement
  Arms: Compression bandage group
Device: Gauze dressing — standard of care gauze dressing placed after total knee replacement
  Arms: Standard gauze group

SUMMARY:
The purpose of this study is to evaluate if applying a compression bandage on the leg alters early outcome following TKA.

The primary objective of this study is to evaluate leg swelling by measuring leg circumference following simultaneous bilateral total knee arthroplasty (TKA) with and without the application of compression bandage.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving elective simultaneous bilateral primary total knee arthroplasty, treated by Rothman physicians at the Thomas Jefferson University Hospital or Rothman Specialty Hospital.

Exclusion Criteria:

* Previous venous thromboembolic event.
* Lymph edema in one or both legs.
* BMI > 40
* Prior surgery (other than arthroscopy)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
swelling of the knee | one day following surgery
  Swelling of the leg will be determined by measuring circumference of the leg

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Morrison, MS, CCRP, Study Director — Rothman Institute
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No